CLINICAL TRIAL: NCT07279766
Title: A Phase 4 Pragmatic, Randomized Trial to Evaluate the Effectiveness of mRNA-1273 Variant-Containing Vaccine Formulation Against Severe Outcomes in Adults Aged 50-64 Years Without Risk Factors for Severe COVID-19
Brief Title: Effectiveness of mRNA-1273 Variant-Containing Vaccine Formulation Against Severe Outcomes in Adults Aged 50-64 Years Without Risk Factors for Severe COVID-19
Acronym: DAN-COVID
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, MSc, MPH, PhD, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAN-COVID; 2025-523841-82-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2025-11-28; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
Keywords: COVID-19; Vaccination; Pragmatic; Registry; Respiratory tract disease; Respiratory; Cardiovascular
MeSH Terms: conditions — COVID-19; Respiratory Tract Diseases | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- mRNA-1273 (Spikevax) (Experimental): COVID-19 vaccine single injection at day 0
  Interventions: Biological: mRNA-1273 (Moderna COVID-19 vaccine)
- No COVID-19 vaccine (control) (No Intervention): Control arm, no COVID-19 vaccine

INTERVENTIONS:
Biological: mRNA-1273 (Moderna COVID-19 vaccine) — For this arm, the current variant formulation of Spikevax (mRNA-1273) vaccine will be used.
  Arms: mRNA-1273 (Spikevax)

SUMMARY:
The purpose of this pragmatic randomized trial is to evaluate the vaccine effectiveness of the COVID-19 vaccine, mRNA-1273, in adults aged 50-64 years without known risk factors for severe COVID-19 infection. Participants will be randomized 1:1 to either COVID-19 vaccine or no COVID-19 vaccine.

DETAILED DESCRIPTION:
The study is a pragmatic, registry-based, open-label, individually randomized trial. The Danish nationwide administrative health registries will be used for data collection including baseline information, follow-up data, and safety monitoring. The study aims to randomize a total of 285,000 participants. Participants will be individually randomized 1:1 to receive either a COVID-19 vaccine or no COVID-19 vaccine. The study is designed to assess the vaccine effectiveness of the COVID-19 vaccine vs. no COVID-19 vaccine on the risk of medically attended COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-64 years
* Informed consent form has been signed and dated

Exclusion Criteria:

* Medical conditions that increase the risk of severe COVID-19, which will be assessed through self-reporting. These medical conditions include:

  1. Asthma
  2. Cancer (excluding non-melanoma skin cancer)
  3. Cardiomyopathies
  4. Cerebrovascular disease
  5. Chronic kidney disease
  6. Chronic lung disease
  7. Cystic Fibrosis
  8. Dementia
  9. Diabetes
  10. Down syndrome
  11. Heart failure
  12. Human Immunodeficiency Virus
  13. Immunosuppressive therapy
  14. Ischemic heart disease
  15. Liver disease
  16. Neurological/neuromuscular disease
  17. Psychiatric disease (psychotic, schizophrenic, schizotypal, depressive, and bipolar (affective) disorders).
  18. Severe obesity (body mass index >35 kg/m2)
  19. Severe substance abuse
  20. Short bowel syndrome
  21. Solid organ transplant or hematological transplant
* Apart from these, there are no specific exclusion criteria for this study

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 285000 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Medically attended COVID-19 | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
  Defined as a positive PCR test for SARS-CoV-2 or hospitalization for COVID-19-related respiratory tract disease

SECONDARY OUTCOMES:
COVID-19-related hospitalization | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
COVID-19-related respiratory tract disease hospitalization | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
COVID-19-related cardio-respiratory disease hospitalization | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
All-cause respiratory tract disease hospitalization | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
All-cause cardio-respiratory hospitalization | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
All-cause lower respiratory tract disease hospitalization | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
All-cause hospitalization | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
COVID-19 death | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
All-cause death | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date

OTHER OUTCOMES:
COVID-19-related hospitalization (alternate definition) | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Laboratory-confirmed COVID-19 | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Total length of hospital stays due to COVID-19-related respiratory tract disease | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Composite of hospitalization for COVID-19 or pneumonia (ICD-10 codes only) | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Hospitalization for any cardiovascular disease | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Hospitalization due to any infectious disease | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Hospitalization requiring mechanical ventilation | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
In-hospital mortality | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Cardio-respiratory mortality | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Respiratory mortality | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Cardiovascular mortality | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Intensive care unit admission | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Laboratory-confirmed COVID-19 hospitalization | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date
Any hospital contact associated with laboratory-confirmed COVID-19 | ≥14 days after initially booked study visit date until 6 months after initially booked study visit date

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, MSc, MPH, PhD, Study Chair — Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (2):
- Denmark (2):
  - Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup
  - Danske Lægers Vaccinations Service, Søborg

IPD SHARING:
Plan to Share IPD: Yes
In this trial, baseline and endpoint data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.
Supporting Information: Study Protocol, SAP